CLINICAL TRIAL: NCT03440918
Title: Prospective, Randomized Controlled Trial to Evaluate the Impact of a Procalcitonin Testing and Treatment Algorithm on Antibiotic Use and Outcomes in the Pediatric Intensive Care Unit
Brief Title: Impact of a Procalcitonin Testing and Treatment Algorithm on Antibiotic Use and Outcomes in the Pediatric Intensive Care Unit
Acronym: ProPICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Sophie Katz, Postdoctoral Fellow, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 170778
Record Dates: First submitted 2018-02-08; First posted 2018-02-22 (Actual); Results first posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Sepsis; Procalcitonin; Antimicrobial Stewardship
Keywords: Infection
MeSH Terms: conditions — Sepsis; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Antimicrobial Stewardship (Active Comparator): Baseline audit of antimicrobial orders with feedback to providers by the antimicrobial stewardship team.
  Interventions: Other: Procalcitonin-Guided Antimicrobial Stewardship; Other: Baseline Antimicrobial Stewardship
- Procalcitonin-Guided Antimicrobial Stewardship (Experimental): In addition to baseline audit of antimicrobial orders, the stewardship team will additionally recommend procalcitonin (PCT) testing and treatment per algorithm. PCT will be used in conjunction with clinical status and exam, and results of radiographic and laboratory studies, to make medical decisions about antibiotic therapy.
  Interventions: Other: Procalcitonin-Guided Antimicrobial Stewardship

INTERVENTIONS:
Other: Procalcitonin-Guided Antimicrobial Stewardship — In addition to baseline audit of antimicrobial orders, the stewardship team will additionally recommend procalcitonin (PCT) testing and treatment per algorithm. PCT will be used in conjunction with clinical status and exam, and results of radiographic and laboratory studies, to make medical decisions about antibiotic therapy.
Other: Baseline Antimicrobial Stewardship — Baseline audit of antimicrobial orders with feedback to providers by the antimicrobial stewardship team.
  Arms: Baseline Antimicrobial Stewardship

SUMMARY:
The timely use of antibiotics can reduce morbidity and mortality associated with bacterial infections, particularly in the intensive care unit setting (ICU). Long courses of antibiotics, however, are associated with the emergence of multi-drug resistant organisms and antibiotic-associated adverse events, such as C. difficile infections. Thus, antibiotic de-escalation is an important goal of antimicrobial stewardship programs.

Procalcitonin (PCT) has been investigated as a biomarker for critically ill adult patients with bacterial infection, particularly pneumonia and sepsis. The proposed project will evaluate whether a PCT testing and treatment algorithm, implemented through daily antimicrobial stewardship audit and feedback, can promote early and safe antibiotic de-escalation in the pediatric ICU.

DETAILED DESCRIPTION:
The timely use of effective antibiotics can markedly reduce the morbidity and mortality associated with bacterial infections, particularly in the intensive care unit (ICU). However, in this setting, much antibiotic use is empiric, and administered to patients with non-bacterial or non-infectious causes of inflammation that do not respond to antibiotics. This widespread empiric use of antibiotics drives the emergence of multi-drug resistant organisms and antibiotic-associated adverse events, such as C. difficile infections. De-escalation of broad-spectrum empiric antibiotics for ICU patients without proven bacterial infections can reduce unnecessary antibiotic use, slow the development of antibiotic resistance, and reduce complications associated with antibiotic therapy. Thus, antibiotic de-escalation is an important goal of antimicrobial stewardship programs. Specific tests and pathways to predict which patients have bacterial infections and those that would benefit from antibiotic therapy would accelerate de-escalation and greatly facilitate antimicrobial stewardship efforts.

Procalcitonin (PCT) has been investigated as a biomarker for critically ill adult patients with bacterial infection, particularly pneumonia and sepsis. Following bacteria-induced activation of monocytes and adherence of monocytes to endothelial surfaces, procalcitonin is expressed and secreted. PCT levels have been shown to rise rapidly and remain elevated during ongoing bacterial infections, and PCT levels are more specific for bacterial infections than CRP or total white blood cell count. PCT rises approximately 4 hours after bacterial exposure, peaks between 12-24 hours, and has a half-life of 24 hours once the infectious stimulus is removed.

In many adult trials investigating PCT-guided algorithms for antibiotic cessation (refer to section 3.0), a high proportion of providers (up to 50%) chose not to follow algorithm guidance for subjects randomized to the PCT-guided group. Thus, although PCT appears to be a useful guide for safe antibiotic de-escalation in the ICU, the ideal method for implementing the test and integrating it into clinical care in order to maximize its impact in the pediatric population is unclear. Notably, none of the prior trials evaluated PCT-associated outcomes in critically ill children nor integrated PCT testing into antimicrobial stewardship activities.

The investigators propose the evaluation of a PCT testing and treatment algorithm on patient outcomes in the pediatric ICU, a setting in which PCT-guided antibiotic de-escalation has not been previously studied.

The proposed project will evaluate whether a procalcitonin (PCT) testing and treatment algorithm, implemented through daily antimicrobial stewardship audit and feedback, can promote early and safe antibiotic de-escalation in the pediatric ICU. The investigators will conduct a pragmatic, prospective randomized controlled trial comparing antimicrobial use and outcomes among children admitted to the ICU who receive either: 1) Routine laboratory testing and treatment with antimicrobial stewardship review (control), or 2) PCT testing and treatment with antimicrobial stewardship review (intervention). In both arms, baseline daily review of antimicrobial management by the stewardship team will occur. In the intervention arm, the stewardship provider also will recommend PCT testing and antibiotic modifications using a PCT-based treatment algorithm. PCT levels will be measured a total of four times in the intervention arm - on enrollment, then daily through day 3 post-randomization and on day 5 post-randomization. This research is not to determine if PCT is a good test; this has already been established and evaluated as part of the FDA approval process. This pragmatic outcomes trial is evaluating if use of the PCT, implemented together with antimicrobial stewardship program oversight, improves the quality of care the investigators can provide for children at Vanderbilt Children's Hospital. The investigators hypothesize that patients in the intervention arm will have shorter duration of antibiotic therapy and similar outcomes, as compared to patients in the control arm.

Specific Aims

1. Compare antimicrobial utilization among children in the ICU who receive standard-of-care testing plus stewardship vs. PCT-based treatment plus stewardship. The investigators will compare days of antibiotic therapy in the first 14 days following randomization between the study arms. The investigators will test the hypothesis that duration of antibiotic therapy will be 2 days shorter in the group with PCT-guided management vs. the group with standard of care testing and treatment.
2. Compare clinical outcomes and safety among children in the ICU who receive standard-of-care testing plus stewardship vs. PCT-based treatment plus stewardship. The investigators will compare mortality, length of stay, recurrence of infection, and antibiotic-associated adverse events (rash, myelosuppression, renal impairment, hepatotoxicity, C. difficile infection) between the study arms. The investigators will test the hypothesis that outcomes and safety will be comparable between the study arms.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or younger
* Prescribed or administered antibiotics in the hospital less than or equal to 24 hours prior to enrollment
* Have parents or legal guardians who provide informed consent
* Provide assent (if > 7 years of age)

Exclusion Criteria:

* Are not prescribed antibiotics in the hospital
* Receive intravenous antibiotics within 7 days prior to identification for study enrollment
* Primary or secondary immune deficiency
* History of malignancy, bone marrow transplant or solid organ transplant
* A diagnosis of cystic fibrosis
* Neonates < 34 weeks gestation
* Patients receiving treatment for endocarditis, osteomyelitis, meningitis, mediastinitis or other invasive infection, for which long duration of antibiotics is needed
* Do not provide informed consent/assent

Ages: 2 Hours to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 271 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2019-05-11 (Actual); Study Completion 2019-05-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ritu Banerjee, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Katz SE, Crook J, Gillon J, Stanford JE, Wang L, Colby JM, Banerjee R. Use of a Procalcitonin-guided Antibiotic Treatment Algorithm in the Pediatric Intensive Care Unit. Pediatr Infect Dis J. 2021 Apr 1;40(4):333-337. doi: 10.1097/INF.0000000000002986. PMID 33181782

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 528 patients in the pediatric ICU were on antibiotics < 1 calandar day and were assessed for eligibility during the study period, February 15, 2018 to April 11, 2019.
  257 were excluded and did not undergo randomization.
Pre-assignment Details: No patients enrolled in the study were excluded before assignment to groups.
Groups:
- Usual Care Antimicrobial Stewardship: Participants received usual care audit of antimicrobial orders with feedback to providers by the antimicrobial stewardship team.
- Procalcitonin-Guided Antimicrobial Stewardship: In addition to usual care audit and feedback of antimicrobial orders, the stewardship team additionally recommended procalcitonin (PCT) testing and treatment per algorithm. PCT was used in conjunction with clinical status and exam, and results of radiographic and laboratory studies, to make medical decisions about antibiotic therapy.
Period: Overall Study
Arm/Group | Usual Care Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Started | 133 | 138
Completed | 133 | 122
Not Completed | 0 | 16
Not completed — Protocol Violation | 0 | 16

BASELINE CHARACTERISTICS:
Population: Modified intention to treat analysis - excludes 1 patient from the procalcitonin arm who underwent cardiac transplant on day 3 after enrollment
Groups:
- Usual Care: Usual Care audit of antimicrobial orders with feedback to providers by the antimicrobial stewardship team.
- Procalcitonin-Guided Antimicrobial Stewardship: In addition to usual care audit and feedback of antimicrobial orders, the stewardship team additionally recommended procalcitonin (PCT) testing and treatment per algorithm. PCT was be used in conjunction with clinical status and exam, and results of radiographic and laboratory studies, to make medical decisions about antibiotic therapy.
- Total: Total of all reporting groups
Arm/Group | Usual Care | Procalcitonin-Guided Antimicrobial Stewardship | Total
Number analyzed (Participants) | 133 | 137 | 270
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 126 | 132 | 258
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 2.3 [0.5 to 8.9] | 1.6 [0.5 to 8.3] | 1.89 [0.49 to 8.63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 57 | 130
  Male | 60 | 80 | 140
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 20 | 30
  Not Hispanic or Latino | 114 | 112 | 226
  Unknown or Not Reported | 9 | 5 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 18 | 36
  White | 103 | 106 | 209
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 12 | 22
Region of Enrollment [Number; unit: participants]
  United States | 133 | 137 | 270
Location at Enrollment [Count of Participants; unit: Participants]
  Medical / Surgical ICU | 111 | 112 | 223
  Cardiac ICU | 22 | 25 | 47
Vasopressor Support [Count of Participants; unit: Participants] | 33 | 27 | 60
Mechanical Ventilation [Count of Participants; unit: Participants] | 61 | 45 | 106
Fever at enrollment [Count of Participants; unit: Participants] | 79 | 61 | 140
Recent surgery [Count of Participants; unit: Participants] | 37 | 24 | 61
Antibiotic Indication [Count of Participants; unit: Participants]
  Sepsis | 51 | 64 | 115
  Pneumonia | 59 | 48 | 107
  Other | 23 | 25 | 48
Final Diagnosis [Count of Participants; unit: Participants]
  Pneumonia | 44 | 41 | 85
  Aspiration pneumonia | 10 | 10 | 20
  Tracheitis | 6 | 12 | 18
  Viral illness | 16 | 12 | 28
  Non-infectious etiology | 23 | 35 | 58
  Other | 34 | 27 | 61

OUTCOME MEASURES:

1. Primary Outcome: Days of Antibiotic Therapy in the First 14 Days Following Randomization
Description: Days of antibiotic therapy a participant receives following randomization will be measured
Time Frame: 14 days
Population: Intention to treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
days | 7.6 [3 to 11.8] | 6.6 [3.1 to 10.9]

2. Secondary Outcome: Duration of Broad-spectrum Antibiotic Therapy
Description: Defined as vancomycin, daptomycin, amikacin, ceftazidime, cefepime, piperacillin/tazobactam, aztreonam, carbapenems
Time Frame: up to14 days
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
days | 0 [0 to 1.8] | 0.086 [0 to 2.6]

3. Secondary Outcome: Number of Patients With an Antibiotic Change
Description: Number of patients with an appropriate antibiotic escalation or de-escalation based on patient's clinical status and available supporting laboratory evidence, or lack thereof, of specific type of infection
Time Frame: up to 14 days
Population: intention to treat (all participants assigned to baseline antimicrobial stewardship or procalcitonin-guided antimicrobial stewardship)
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
Participants | 111 | 108

4. Secondary Outcome: 30-day Mortality
Description: All-cause mortality
Time Frame: up to 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
Participants | 4 | 3

5. Secondary Outcome: Re-initiation of Antibiotics for a Bacterial Infection
Description: Re-initiation of any antibiotic for a proven or suspected bacterial infection
Time Frame: up to 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
Participants | NA — Insufficient number of participants with events | NA — Insufficient number of participants with events

6. Secondary Outcome: Length of Intensive Care Unit Stay
Description: Hospital days spent in the intensive care unit
Time Frame: up to 14 days
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
days | 2 [1 to 5] | 2 [1 to 6]

7. Secondary Outcome: Length of Overall Hospital Stay
Description: Hospital days admitted to the hospital
Time Frame: Until hospital discharge, an average of 7 days
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
days | 7 [3 to 12] | 6 [4 to 14]

8. Secondary Outcome: Ventilator Days
Description: Days spent using invasive ventilation methods (not including supplementary oxygen via nasal cannula or Vapotherm support)
Time Frame: up to 14 days
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
days | 3.9 [2.4 to 6.1] | 4.4 [2.5 to 11.1]

9. Secondary Outcome: Number of Participants With Antibiotic-associated Complications
Description: Antibiotic-associated complications including rash, neutropenia, thrombocytopenia, acute kidney injury [defined as increase in serum creatinine > 0.3 mg per dL or > 1.5-fold from baseline, or urine output < 0.5 mL per kg per hour for more than six hours], hepatotoxicity [defined as > 2-fold increase in alanine aminotransferase, ALT, or conjugated bilirubin], or C. difficile infection will be recorded
Time Frame: up to 14 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
Participants | 2 | 3

10. Secondary Outcome: Infection With a Multi-drug Resistant Organism
Description: Identification/growth of a multi-drug resistant organism from a sterile culture site. Multi-drug resistant organisms will be defined as methicillin-resistant S. aureus, vancomycin-resistant Enterococcus, 3rd generation cephalosporin non-susceptible Enterobacteriaceae, multi-drug resistant Pseudomonas aeruginosa [resistant to aminoglycosides, cephalosporins, floroquinolones and carbepenems], carbepenem-resistant Acinetobacter, and Candida spp obtained from otherwise sterile sites [i.e. blood or urine cultures]
Time Frame: up to 30 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
Participants | 1 | 2

11. Secondary Outcome: Antibiotic Cost
Description: Cost of antibiotic course will be obtained from hospital billing data
Time Frame: up to 14 days
Population: as for outcome 3
Measure: Number; unit: dollars
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
dollars | NA — data not collected | NA — data not collected

12. Secondary Outcome: Number of Participants Whose Provider Adhered to the Procalcitonin-guided Algorithm
Description: Rate of clinical provider compliance with adherence to suggested antibiotic escalation or de-escalation made by the antimicrobial stewardship team based on procalcitonin levels will be tracked
Time Frame: up to 5 days
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
Number analyzed (Participants) | 133 | 137
Participants | 123 | 121

ADVERSE EVENTS:
Time Frame: 30 days
Description: Adverse events were collected as part of the safety outcomes. Providers were able to overrule antibiotic stewardship recommendations.
Arm/Group | Baseline Antimicrobial Stewardship | Procalcitonin-Guided Antimicrobial Stewardship
All-Cause Mortality (participants affected / at risk) | 4/133 | 3/137
Serious Adverse Events (participants affected / at risk) | 0/133 | 0/137
Other Adverse Events (participants affected / at risk) | 0/133 | 0/137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT03440918/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/18/NCT03440918/SAP_001.pdf